CLINICAL TRIAL: NCT01361230
Title: PILOT STUDY: A Randomized Controlled Trial of Intensive Care Management of Sedation Using Patient Responsiveness in Critical Care IMPROVE Critical Care Study Pilot
Brief Title: IMPROVE Critical Care Study (Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Professor Timothy Walsh, Principal investigator, Royal Infirmary of Edinburgh (Great Britain)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DOC0676170
Record Dates: First submitted 2010-04-19; First posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Sedated ICU Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocol (Experimental): Using sedation monitoring and protocol
  Interventions: Device: "Sedation Trial Monitor" is the name of the device used.
- Control (No Intervention): Standard practice

INTERVENTIONS:
Device: "Sedation Trial Monitor" is the name of the device used. — This is a pilot unblinded randomised controlled trial comparing sedation management using responsiveness (new intervention) with usual care (control group).
  Arms: Protocol

SUMMARY:
The Pilot Clinical Investigation planned is a prospective, unblinded randomized pilot trial comparing sedation management using a protocol based on responsiveness with standard sedation management. The hypothesis is that responsiveness will improve a range of patient-based and economic outcomes, including the duration of mechanical ventilation and duration of coma in the ICU. The purpose of the pilot study is to gather information for designing a full study that might show the validity of the outcome hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Patients mechanically ventilated via an endotracheal tube and receiving intravenous sedation with a hypnotic agent (midazolam or other benzodiazepine) or propofol by continuous infusion.

Exclusion Criteria:

* Primary intracerebral disorder (includes cardiac arrest with probable hypoxic brain injury; intrac-ranial haemorrhage; head injury causing reduced conscious level prior to intubation)
* Patient who is already awake at the time of enrolment defined as RASS ³ -1
* Age <16 years
* Patient not expected to survive the next 24 hours
* Patient receiving long term ventilation prior to ICU admission
* Patient with a long term tracheostomy prior to ICU admission
* Patient transferred sedated and mechanically ventilated from another ICU unless recruitment is possible within 24 hours of first ICU admission
* Patient receiving continuous neuromuscular blocking agent at the time of screening for enrolment
* Previously enrolled in the trial during a separate ICU admission during this hospital stay
* Status epilepticus
* Confirmed meningitis or encephalitis at the time of screening for enrolment
* Chronic neurological disease interfering with normal neuromuscular function, e.g. motor neurone disease, Guillain-Barre syndrome or inherited neuromyopathies

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Proportion of time spent with low responsiveness (red colour code) during the first 48 hours in the ICU | 8 month period
  The main purpose in the statistical analysis is not to test the statistical significance of the differences but to provide descriptive statistics for the full outcome study plan.

SECONDARY OUTCOMES:
Proportion of time spent with RASS score -4/-5 during the first 48 hours in the ICU. | 8 months
  The main purpose in the statistical analysis is not to test the statistical significance of the differences but to provide descriptive statistics for the full outcome study plan.

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Uutela, PhD, Study Director — GEHC; Timothy Walsh, PhD MD, Principal Investigator — Royal Infirmary of Edinburgh
Locations (1):
- Royal Infirmary Edinburgh (Great Britain) ward 118, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Kaila M, Everingham K, Lapinlampi P, Peltola P, Sarkela MO, Uutela K, Walsh TS. A randomized controlled proof-of-concept trial of early sedation management using Responsiveness Index monitoring in mechanically ventilated critically ill patients. Crit Care. 2015 Sep 11;19(1):333. doi: 10.1186/s13054-015-1043-1. PMID 26370687